CLINICAL TRIAL: NCT04902430
Title: Evaluation of the Rate of En-masse Retraction in Orthodontic Patients With Maxillary Protrusion Using Friction Versus Frictionless Mechanics: A Randomized Clinical Trial
Brief Title: Evaluation of the Rate of En-masse Retraction in Orthodontic Patients With Maxillary Protrusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Leena Alaa Shibl, Principle Investigator, Future University in Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUE.REC (8)/6-2019
Record Dates: First submitted 2021-05-12; First posted 2021-05-26 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Bimaxillary Protrusion
Keywords: En-masse Retraction; Friction; Fricitionless; Lateral Cephalometric; Rate; Dental Models

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Only the outcome assessors will be blind. The patients name will be sealed from pre and post radiographs and study models. Then two assessors will carry out, blindly and independently, the measurements and analysis of the study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- En-Masse Retraction using sliding mechanics (Friction) (Experimental): 6 anterior teeth (en-Masse) retracted using a crimpable hook distal to the upper lateral incisor and a power chain
  Interventions: Procedure: Power chain and Crimpable hook for En-Masse Retraction
- En-Masse Retraction using segmental mechanics (Frictionless) (Experimental): 6 anterior teeth (en-Masse) retracted using a T- loop
  Interventions: Procedure: T- Loop

INTERVENTIONS:
Procedure: Power chain and Crimpable hook for En-Masse Retraction — Retraction will start on a 0.017"x0.025" Stainless steel wire using elastomeric chain (force applied will be 212 g per side) extending between the crimpable hooks and the miniscrew
  Arms: En-Masse Retraction using sliding mechanics (Friction)
Procedure: T- Loop — Closing retraction T-loops will be fabricated using 0.017 x 0.025 TMA wire. The loop will be positioned halfway the extraction space and the canine
  Arms: En-Masse Retraction using segmental mechanics (Frictionless)

SUMMARY:
There's a scarcity in literature concerning en-masse retraction and its effect on the rate of tooth movement. The purpose of this study is to determine, In orthodontic patients with maxillary protrusion, which form of mechanics in en-masse retraction offers a faster rate of retraction; Friction or Frictionless Mechanics.

DETAILED DESCRIPTION:
The en-masse technique can be done in one of two ways: through friction or frictionless mechanics. Both are viable options, but, ideally, we want to retract and complete the orthodontic treatment as quickly as possible, in order to decrease the negative effects that may occur during treatment. Which of these mechanics results in a decreased treatment time is still up for debate.

ELIGIBILITY:
Inclusion Criteria:

* Adults and Adolescent patients (both genders)
* Age range (14-24)
* Patients with maxillary protrusion requiring first premolars extraction (Bimaxillary Protrusion or Class II division 1 cases).
* Patients with fully erupted permanent teeth (not necessarily including the third molar).
* Cases requiring maximum anchorage during retraction.
* Good general and oral health

Exclusion Criteria:

* Patients suffering from any systemic diseases interfering with tooth movement.
* Patients with extracted or missing permanent teeth. (except for third molars).
* Patients with badly decayed teeth.
* Patients with any parafunctional habits (i.e. Bruxism, tongue thrusting, mouth breathing, etc…).
* Patients with previous orthodontic treatment

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2020-12-29 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2022-08-12 (Actual)

PRIMARY OUTCOMES:
Retraction Rate | From pre to post retraction (an average of 6 - 8 months)
  The antero-posterior movement of anterior teeth and first molars will be assessed by measuring the digitilized study models taken of the patients monthly (measured in mm)

SECONDARY OUTCOMES:
Anchorage Loss | From pre to post retraction (an average of 6 - 8 months)
  Digitilized dental models taken before and after the completion of retraction will be measured by identifying landmarks and reference lines and planes (measured in mm)
Molar Rotation | From pre to post retraction (an average of 6 - 8 months)
  Study models that are taken pre and post retraction (then digitilized) will be used to assess the rotation of the maxillary first molars in relation to a reference line (measurement of the angles in degrees)
Pain of intervention | From pre to post retraction/intervention (an average of 6 - 8 months)
  Each patient will fill a questionnaire regarding his treatment experience in a VAS scoring from 1-10
Anterior teeth torque, extrusion/intrusion | From pre to post retraction (an average of 6 - 8 months)
  The principle investigator will examine pre and post lateral cephalometric radiographs in relation to lines and reference planes (measurements in degrees and mm)

CONTACTS AND LOCATIONS:
Overall Officials: Yehia Mostafa, Professor and Chairman, Study Director — Future University in Egypt
Locations (1):
- Future University in Egypt, New Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after publication

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-12-01): https://cdn.clinicaltrials.gov/large-docs/30/NCT04902430/Prot_SAP_000.pdf
  • Informed Consent Form (2019-12-01): https://cdn.clinicaltrials.gov/large-docs/30/NCT04902430/ICF_001.pdf